CLINICAL TRIAL: NCT00878995
Title: Nutrition and Anabolic Interventions in Squamous Cell Carcinoma
Brief Title: Testosterone for Treating Cachexia in Patients With Squamous Cell Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 06-073/10-207; R01CA127971 (NIH); CDR0000629579; GCRC#724/819
Record Dates: First submitted 2009-04-08; First posted 2009-04-09 (Estimated); Results first posted 2018-03-12 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Cachexia; Squamous Cell Carcinoma
Keywords: stage IIB cervical cancer; stage III cervical cancer; recurrent cervical cancer; cachexia; advanced head/neck carcinoma; recurrent head/neck carcinoma
MeSH Terms: conditions — Cachexia; Carcinoma, Squamous Cell; Uterine Cervical Neoplasms | interventions — testosterone enanthate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care Therapy + Placebo Testosterone (Placebo Comparator): Patients receive standard of care chemotherapy and/or radiation plus placebo testosterone intramuscularly (IM) weekly for 7 weeks.
  Interventions: Drug: Placebo Testosterone
- Standard of Care Therapy + Testosterone (Active Comparator): Patients receive standard of care chemotherapy and/or radiation plus testosterone (Testosterone Enanthate 100mg/ml) intramuscularly (IM) weekly for 7 weeks.
  Interventions: Drug: Testosterone Enanthate 100 MG/ML

INTERVENTIONS:
Drug: Placebo Testosterone — Placebo (Saline) Testosterone given IM once per week.
  Arms: Standard of Care Therapy + Placebo Testosterone
Drug: Testosterone Enanthate 100 MG/ML — Testosterone Enanthate 100mg/ml given once per week IM.
  Arms: Standard of Care Therapy + Testosterone

SUMMARY:
RATIONALE: Testosterone may lessen weight loss and improve muscle size and strength in patients with cachexia caused by cancer.

PURPOSE: This randomized phase I trial is studying whether testosterone administered during standard of care chemotherapy and/or radiation works by helping patients with squamous cell carcinoma to maintain their body weight and muscle size and strength during treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the effect of testosterone therapy on lean body mass and muscle strength in patients with advanced or recurrent squamous cell carcinoma.
* To determine the testosterone therapy on inflammatory biomarkers in patients with advanced or recurrent squamous cell carcinoma.

OUTLINE: Patients are stratified according to age and disease stage. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive standard of care chemotherapy and/or radiation and placebo testosterone intramuscularly (IM) weekly for 7 weeks.
* Arm II: Patients receive standard of care chemotherapy and/or radiation and testosterone IM weekly for 7 weeks.

Patients undergo dual energy x-ray absorptiometry, muscle strength tests, stable isotope metabolic studies, indirect calorimetry studies, and assessment of their physical activity level, and nutritional counseling. Patients also complete mood, fatigue, and quality-of-life questionnaires.

Blood, muscle tissue, and urine samples are collected periodically for laboratory studies. Samples are analyzed for serum inflammatory biomarkers and inflammatory cytokines by immunoassay.

After completion of study treatment, patients are followed periodically for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of advanced (stage IIB, IIIA, or IIIB) or recurrent squamous cell carcinoma
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Mini Mental State Examination score > 23

Exclusion Criteria:

* Pregnancy
* Evidence of hepatitis as indicated by a 3-fold increase in 2 out of 3 liver enzymes
* Significant liver, renal, or heart disease
* Diabetes mellitus or other untreated endocrine disease
* Polycystic ovary syndrome and/or hyperthecosis
* Androgen secreting tumors of the ovary and adrenal or any ovarian tumors (e.g., Sertoli- Leydig cell tumor)
* Non-classical adrenal hyperplasia
* Cushing's syndrome
* Glucocorticoid resistance
* Hyperprolactinoma or hypothyroidism
* Lactose intolerance
* Alcohol or drug abuse
* Recent treatment (within 3 months) with anabolic steroids
* Ongoing anticoagulant therapy
* Any other circumstance that would preclude study participation, in the opinion of the principal investigator or study physician

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2009-06-03 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melinda Sheffield-Moore, PhD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

REFERENCES:
- [Derived] Scott JM, Dillon EL, Kinsky M, Chamberlain A, McCammon S, Jupiter D, Willis M, Hatch S, Richardson G, Danesi C, Randolph K, Durham W, Wright T, Urban R, Sheffield-Moore M. Effects of adjunct testosterone on cardiac morphology and function in advanced cancers: an ancillary analysis of a randomized controlled trial. BMC Cancer. 2019 Aug 7;19(1):778. doi: 10.1186/s12885-019-6006-5. PMID 31391011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited via UTMB Oncology, Radiation Oncology, and ENT clinics by study physicians.
Pre-assignment Details: Subjects began study before beginning chemotherapy and/or radiation therapy. 28 subjects enrolled total. 4 subjects withdrew before beginning the study.
Groups:
- Arm I: Standard of Care Therapy + Placebo Testosterone: Patients receive standard of care chemotherapy and/or radiation plus placebo testosterone intramuscularly (IM) weekly for 7 weeks.
  Standard of Care Chemotherapy and/or Radiation plus Placebo (Saline) Testosterone: Standard of Care Chemotherapy and/or Radiation plus Placebo (Saline) Testosterone
- Arm II: Standard of Care Therapy + Testosterone: Patients receive standard of care chemotherapy and/or radiation plus testosterone intramuscularly (IM) weekly for 7 weeks.
  Arm II: Standard of Care Chemotherapy and/or Radiation plus Testosterone Enanthate: Arm II: Standard of Care Chemotherapy and/or Radiation plus Testosterone Enanthate
Period: Baseline Study - Midpoint Study
Arm/Group | Arm I: Standard of Care Therapy + Placebo Testosterone | Arm II: Standard of Care Therapy + Testosterone
Started | 12 | 12
Baseline Study | 12 | 12
Completed | 12 | 10 (2 subjects dropped after the baseline study. They decided to seek treatment closer to home.)
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2
Period: Midpoint Study - Post Study
Arm/Group | Arm I: Standard of Care Therapy + Placebo Testosterone | Arm II: Standard of Care Therapy + Testosterone
Started | 12 | 10
Completed | 12 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I: Standard of Care Therapy + Placebo Testosterone | Arm II: Standard of Care Therapy + Testosterone | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (7.97) | 48.66 (12.26) | 51.44 (10.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 14
  Male | 7 | 3 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 10 | 11 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 10 | 10 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Lean Body Mass as Measured by Dual Energy X-ray Absorptiometry (DEXA) From Baseline to 7 Weeks.
Description: Total Lean Body Mass was measured on a GE Lunar iDEXA at baseline and 7 weeks. Percent change from baseline to 7 weeks is reported.
Time Frame: 7 weeks
Population: Reporting data for the 22 completing subjects only, since this data is reported as change over time.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Arm I: Standard of Care Therapy + Placebo Testosterone | Arm II: Standard of Care Therapy + Testosterone
Number analyzed (Participants) | 12 | 10
Percent change | -3.31 (6.34) | 1.42 (7.25)

2. Secondary Outcome: Maximum Peak Isometric Leg Strength as Measured by Biodex Pro4 at Baseline
Description: Peak isometric strength is measured on a Biodex System 4 Pro. This test is isolated to the quadricep muscle of one leg. Isometric test is performed at 90 degrees with 5 seconds of force production for each contraction. There was 1 set of 3 contractions at 100% force performed.
Time Frame: Baseline
Population: 24 subjects started the study but only 20 subjects were able to complete this outcome measure due to problems relating to their cancer.
Measure: Mean (Standard Deviation); unit: Newton-Meters
Arm/Group | Arm I: Standard of Care Therapy + Placebo Testosterone | Arm II: Standard of Care Therapy + Testosterone
Number analyzed (Participants) | 11 | 9
Newton-Meters | 81.77 (42.58) | 122.50 (70.78)

3. Secondary Outcome: Maximum Peak Isometric Leg Strength as Measured by Biodex Pro 4 at 7 Weeks.
Description: Peak isometric strength is measured on a Biodex System 4 Pro. This test is isolated to the quadricep muscle of one leg. Isometric test is performed at 90 degrees with 5 seconds of force production for each contraction. There was 1 set of 3 contractions at 100% force performed. This outcome was measured after 7 weeks of treatment with study medication.
Time Frame: 7 weeks
Population: Only 15 subjects were able to complete this outcome measure at this time point due to problems related to their cancer.
Measure: Mean (Standard Deviation); unit: Newton-Meters
Arm/Group | Arm I: Standard of Care Therapy + Placebo Testosterone | Arm II: Standard of Care Therapy + Testosterone
Number analyzed (Participants) | 6 | 9
Newton-Meters | 76.75 (25.22) | 118.26 (62.26)

4. Secondary Outcome: Maximum Peak Isokinetic Leg Strength as Measured by Biodex Pro 4 at Baseline.
Description: Isokinetic strength (knee extension) is measured on a Biodex System Pro 4 within a 75 degree range of motion. Subjects performed concentric contractions at a fixed speed of 120 degree/sec. 1 set of 3 contractions were performed at 100% force.
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Watts
Arm/Group | Arm I: Standard of Care Therapy + Placebo Testosterone | Arm II: Standard of Care Therapy + Testosterone
Number analyzed (Participants) | 11 | 9
Watts | 137.60 (86.77) | 169.0 (99.71)

5. Secondary Outcome: Maximum Peak Isokinetic Leg Extension as Measured by Biodex Pro 4 at 7 Weeks
Description: Isokinetic strength (knee extension) is measured on a Biodex System Pro 4 within a 75 degree range of motion set at a fixed speed of 120 degree/sec.
Time Frame: 7 weeks
Population: Only 15 subjects were able to complete this outcome measure at this time point due to problems related to their cancer.
Measure: Mean (Standard Deviation); unit: Watts
Arm/Group | Arm I: Standard of Care Therapy + Placebo Testosterone | Arm II: Standard of Care Therapy + Testosterone
Number analyzed (Participants) | 6 | 9
Watts | 126.93 (57.05) | 157.90 (84.49)

6. Secondary Outcome: Body Weight as Measured by Scale at Baseline
Description: Body weight in kilograms as measured by a scale at the baseline visit.
Time Frame: Baseline
Population: 24 subjects began the study. Each subjects was able to complete this outcome measure at the baseline time point.
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Arm I: Standard of Care Therapy + Placebo Testosterone | Arm II: Standard of Care Therapy + Testosterone
Number analyzed (Participants) | 12 | 12
Kilograms | 65.98 (25.49) | 63.11 (17.24)

7. Secondary Outcome: Body Weight as Measured by Scale at 7 Weeks.
Description: Body Weight in kilograms as measured on a scale after 7 weeks of treatment with the study medication.
Time Frame: 7 weeks
Population: 22 subjects completed this outcome measure at the 7 week time point. 24 subjects started the study, 2 subjects dis-enrolled after the baseline visit.
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Arm I: Standard of Care Therapy + Placebo Testosterone | Arm II: Standard of Care Therapy + Testosterone
Number analyzed (Participants) | 12 | 10
Kilograms | 63.93 (24.79) | 62.59 (17.83)

8. Secondary Outcome: Energy Expenditure Reported as Kcal/Day as Measured by Indirect Calorimetry at Baseline
Description: Energy expenditure and substrate oxidation as measured by indirect calorimetry using expired gases collected and analyzed for oxygen and carbon dioxide concentrations. 30 minutes of sampling was performed, the last 25 minutes were averaged to calculate mean Kcal/day values.
Time Frame: Baseline
Population: 24 subjects completed this outcome measure at the baseline visit.
Measure: Mean (Standard Deviation); unit: kilo-calories per day
Arm/Group | Arm I: Standard of Care Therapy + Placebo Testosterone | Arm II: Standard of Care Therapy + Testosterone
Number analyzed (Participants) | 12 | 12
kilo-calories per day | 1329.20 (359.94) | 1310.81 (398.16)

9. Secondary Outcome: Energy Expenditure Reported as Kcal/Day as Measured by Indirect Calorimetry at 7 Weeks
Description: as for outcome 8
Time Frame: 7 weeks
Population: Only 19 subjects were able to complete this outcome measure at this time point due to problems related to their cancer.
Measure: Mean (Standard Deviation); unit: kilo-calories per day
Arm/Group | Arm I: Standard of Care Therapy + Placebo Testosterone | Arm II: Standard of Care Therapy + Testosterone
Number analyzed (Participants) | 9 | 10
kilo-calories per day | 1338.10 (281.77) | 1260.98 (222.32)

10. Secondary Outcome: Physical Activity Levels as Measured by the ActiGraph Accelerometer
Description: Physical activity is reported as % time sedentary for the entire 7 week study.
Time Frame: through study completion,up to 7 weeks
Population: Data from only 12 subjects is presented due to a compliance issue with wearing the activity monitoring belts. A threshold was set to determine if subject was wearing the belt as directed.
Measure: Mean (Standard Deviation); unit: % time sedentary
Arm/Group | Arm I: Standard of Care Therapy + Placebo Testosterone | Arm II: Standard of Care Therapy + Testosterone
Number analyzed (Participants) | 3 | 9
% time sedentary | 73.55 (15.78) | 74.74 (9.44)

11. Secondary Outcome: Concentration of Cytokine Granulocyte-macrophage Colony-stimulating Factor (GM-CSF) in Blood as Measured by Immunoassay at Baseline
Description: Concentration of cytokine granulocyte-macrophage colony-stimulating factor (GM-CSF) in blood as measured using Millipore Multiplex Human Cytokine Panel assay.
Time Frame: Baseline
Population: Blood was collected for this outcome from only 18 subjects.
Measure: Mean (Standard Deviation); unit: picogram/milliliter
Arm/Group | Arm I: Standard of Care Therapy + Placebo Testosterone | Arm II: Standard of Care Therapy + Testosterone
Number analyzed (Participants) | 11 | 7
picogram/milliliter | 67.02 (67.13) | 260.69 (251.07)

12. Secondary Outcome: Concentration of Cytokine Granulocyte-macrophage Colony-stimulating Factor (GM-CSF) in Blood as Measured by Immunoassay at 7 Weeks
Description: as for outcome 11
Time Frame: 7 weeks
Population: Blood was collected for this outcome from only 18 subjects.
Measure: Mean (Standard Deviation); unit: picogram/milliliter
Arm/Group | Arm I: Standard of Care Therapy + Placebo Testosterone | Arm II: Standard of Care Therapy + Testosterone
Number analyzed (Participants) | 11 | 7
picogram/milliliter | 64.15 (50.36) | 191.17 (206.32)

13. Secondary Outcome: Concentration of Cytokine Interferon-gamma (IFN Gamma) in Blood as Measured by Immunoassay at Baseline.
Description: Concentration of cytokine Interferon-gamma (IFN gamma) in blood as measured using Millipore Multiplex Human Cytokine Panel assay.
Time Frame: baseline
Population: Blood was collected for this outcome from only 18 subjects.
Measure: Mean (Standard Deviation); unit: picogram/milliliter
Arm/Group | Arm I: Standard of Care Therapy + Placebo Testosterone | Arm II: Standard of Care Therapy + Testosterone
Number analyzed (Participants) | 11 | 7
picogram/milliliter | 21.62 (15.61) | 15.71 (7.89)

14. Secondary Outcome: Concentration of Cytokine Interferon-gamma (IFN Gamma) in Blood as Measured by Immunoassay at 7 Weeks
Description: as for outcome 13
Time Frame: 7 weeks
Population: Blood was collected for this outcome from only 18 subjects.
Measure: Mean (Standard Deviation); unit: picogram/milliliter
Arm/Group | Arm I: Standard of Care Therapy + Placebo Testosterone | Arm II: Standard of Care Therapy + Testosterone
Number analyzed (Participants) | 11 | 7
picogram/milliliter | 20.63 (13.01) | 11.66 (8.17)

15. Secondary Outcome: Concentration of Cytokine Interleukin 1 Beta (IL-1B) in Blood as Measured by Immunoassay at Baseline.
Description: Concentration of cytokine Interleukin 1 beta (IL-1B) in blood as measured using Millipore Multiplex Human Cytokine Panel assay.
Time Frame: Baseline
Population: Blood was collected for this outcome from only 18 subjects.
Measure: Mean (Standard Deviation); unit: picogram/milliliter
Arm/Group | Arm I: Standard of Care Therapy + Placebo Testosterone | Arm II: Standard of Care Therapy + Testosterone
Number analyzed (Participants) | 11 | 7
picogram/milliliter | 3.11 (1.95) | 1.98 (0.60)

16. Secondary Outcome: Concentration of Cytokine Interleukin 1 Beta (IL-1B) in Blood as Measured by Immunoassay at 7 Weeks.
Description: as for outcome 15
Time Frame: 7 weeks
Population: Blood was collected for this outcome from only 18 subjects.
Measure: Mean (Standard Deviation); unit: picogram/milliliter
Arm/Group | Arm I: Standard of Care Therapy + Placebo Testosterone | Arm II: Standard of Care Therapy + Testosterone
Number analyzed (Participants) | 11 | 7
picogram/milliliter | 2.13 (2.02) | 1.71 (1.01)

17. Secondary Outcome: Concentration of Cytokine Interleukin 2 (IL-2) in Blood as Measured by Immunoassay at Baseline.
Description: Concentration of cytokine Interleukin 2 (IL-2) in blood as measured using Millipore Multiplex Human Cytokine Panel assay.
Time Frame: baseline
Population: Blood was collected for this outcome from only 18 subjects.
Measure: Mean (Standard Deviation); unit: picogram/milliliter
Arm/Group | Arm I: Standard of Care Therapy + Placebo Testosterone | Arm II: Standard of Care Therapy + Testosterone
Number analyzed (Participants) | 11 | 7
picogram/milliliter | 3.62 (2.87) | 3.92 (2.33)

18. Secondary Outcome: Concentration of Cytokine Interleukin 2 (IL-2) in Blood as Measured by Immunoassay at 7 Weeks.
Description: as for outcome 17
Time Frame: 7 weeks
Population: Blood was collected for this outcome from only 18 subjects.
Measure: Mean (Standard Deviation); unit: picogram/milliliter
Arm/Group | Arm I: Standard of Care Therapy + Placebo Testosterone | Arm II: Standard of Care Therapy + Testosterone
Number analyzed (Participants) | 11 | 7
picogram/milliliter | 3.02 (2.67) | 2.39 (1.43)

19. Secondary Outcome: Concentration of Cytokine Interleukin 4 (IL-4) in Blood as Measured by Immunoassay at Baseline.
Description: Concentration of cytokine Interleukin 4 (IL-4) in blood as measured using Millipore Multiplex Human Cytokine Panel assay.
Time Frame: baseline
Population: Blood was collected for this outcome from only 18 subjects.
Measure: Mean (Standard Deviation); unit: picogram/milliliter
Arm/Group | Arm I: Standard of Care Therapy + Placebo Testosterone | Arm II: Standard of Care Therapy + Testosterone
Number analyzed (Participants) | 11 | 7
picogram/milliliter | 4.30 (4.70) | 3.13 (2.64)

20. Secondary Outcome: Concentration of Cytokine Interleukin 4 (IL-4) in Blood as Measured by Immunoassay at 7 Weeks.
Description: as for outcome 19
Time Frame: 7 weeks
Population: Blood was collected for this outcome from only 18 subjects.
Measure: Mean (Standard Deviation); unit: picogram/milliliter
Arm/Group | Arm I: Standard of Care Therapy + Placebo Testosterone | Arm II: Standard of Care Therapy + Testosterone
Number analyzed (Participants) | 11 | 7
picogram/milliliter | 10.48 (24.43) | 2.35 (2.85)

21. Secondary Outcome: Concentration of Cytokine Interleukin 5 (IL-5) in Blood as Measured by Immunoassay at Baseline.
Description: Concentration of cytokine Interleukin 5 (IL-5) in blood as measured using Millipore Multiplex Human Cytokine Panel assay.
Time Frame: Baseline
Population: Blood was collected for this outcome from only 18 subjects.
Measure: Mean (Standard Deviation); unit: picogram/milliliter
Arm/Group | Arm I: Standard of Care Therapy + Placebo Testosterone | Arm II: Standard of Care Therapy + Testosterone
Number analyzed (Participants) | 11 | 7
picogram/milliliter | 3.02 (2.22) | 14.56 (26.29)

22. Secondary Outcome: Concentration of Cytokine Interleukin 5 (IL-5) in Blood as Measured by Immunoassay at 7 Weeks.
Description: as for outcome 21
Time Frame: 7 weeks
Population: Blood was collected for this outcome from only 18 subjects.
Measure: Mean (Standard Deviation); unit: picogram/milliliter
Arm/Group | Arm I: Standard of Care Therapy + Placebo Testosterone | Arm II: Standard of Care Therapy + Testosterone
Number analyzed (Participants) | 11 | 7
picogram/milliliter | 3.13 (1.98) | 12.62 (24.71)

23. Secondary Outcome: Concentration of Cytokine Interleukin 6 (IL-6) in Blood as Measured by Immunoassay at Baseline.
Description: Concentration of cytokine Interleukin 6 (IL-6) in blood as measured using Millipore Multiplex Human Cytokine Panel assay.
Time Frame: baseline
Population: Blood was collected for this outcome from only 18 subjects.
Measure: Mean (Standard Deviation); unit: picogram/milliliter
Arm/Group | Arm I: Standard of Care Therapy + Placebo Testosterone | Arm II: Standard of Care Therapy + Testosterone
Number analyzed (Participants) | 11 | 7
picogram/milliliter | 11.04 (15.94) | 43.99 (59.45)

24. Secondary Outcome: Concentration of Cytokine Interleukin 6 (IL-6) in Blood as Measured by Immunoassay at 7 Weeks.
Description: as for outcome 23
Time Frame: 7 weeks
Population: Blood was collected for this outcome from only 18 subjects.
Measure: Mean (Standard Deviation); unit: picogram/milliliter
Arm/Group | Arm I: Standard of Care Therapy + Placebo Testosterone | Arm II: Standard of Care Therapy + Testosterone
Number analyzed (Participants) | 11 | 7
picogram/milliliter | 8.89 (5.48) | 23.09 (36.54)

25. Secondary Outcome: Concentration of Cytokine Interleukin 7 (IL-7) in Blood as Measured by Immunoassay at Baseline.
Description: Concentration of cytokine Interleukin 7 (IL-7) in blood as measured using Millipore Multiplex Human Cytokine Panel assay.
Time Frame: Baseline
Population: Blood was collected for this outcome from only 18 subjects.
Measure: Mean (Standard Deviation); unit: picogram/milliliter
Arm/Group | Arm I: Standard of Care Therapy + Placebo Testosterone | Arm II: Standard of Care Therapy + Testosterone
Number analyzed (Participants) | 11 | 7
picogram/milliliter | 6.57 (2.49) | 21.61 (36.35)

26. Secondary Outcome: Concentration of Cytokine Interleukin 7 (IL-7) in Blood as Measured by Immunoassay at 7 Weeks.
Description: as for outcome 25
Time Frame: 7 weeks
Population: Blood was collected for this outcome from only 18 subjects.
Measure: Mean (Standard Deviation); unit: picogram/milliliter
Arm/Group | Arm I: Standard of Care Therapy + Placebo Testosterone | Arm II: Standard of Care Therapy + Testosterone
Number analyzed (Participants) | 11 | 7
picogram/milliliter | 9.97 (7.35) | 18.16 (25.88)

27. Secondary Outcome: Concentration of Cytokine Interleukin 8 (IL-8) in Blood as Measured by Immunoassay at Baseline.
Description: Concentration of cytokine Interleukin 8 (IL-8) in blood as measured using Millipore Multiplex Human Cytokine Panel assay.
Time Frame: Baseline
Population: Blood was collected for this outcome from only 18 subjects.
Measure: Mean (Standard Deviation); unit: picogram/milliliter
Arm/Group | Arm I: Standard of Care Therapy + Placebo Testosterone | Arm II: Standard of Care Therapy + Testosterone
Number analyzed (Participants) | 11 | 7
picogram/milliliter | 14.57 (9.93) | 16.62 (8.20)

28. Secondary Outcome: Concentration of Cytokine Interleukin 8 (IL-8) in Blood as Measured by Immunoassay at 7 Weeks.
Description: as for outcome 27
Time Frame: 7 weeks
Population: Blood was collected for this outcome from only 18 subjects.
Measure: Mean (Standard Deviation); unit: picogram/milliliter
Arm/Group | Arm I: Standard of Care Therapy + Placebo Testosterone | Arm II: Standard of Care Therapy + Testosterone
Number analyzed (Participants) | 11 | 7
picogram/milliliter | 11.45 (5.90) | 12.34 (7.82)

29. Secondary Outcome: Concentration of Cytokine Interleukin 10 (IL-10) in Blood as Measured by Immunoassay at Baseline.
Description: Concentration of cytokine Interleukin 10 (IL-10) in blood as measured using Millipore Multiplex Human Cytokine Panel assay.
Time Frame: baseline
Population: Blood was collected for this outcome from only 18 subjects.
Measure: Mean (Standard Deviation); unit: picogram/milliliter
Arm/Group | Arm I: Standard of Care Therapy + Placebo Testosterone | Arm II: Standard of Care Therapy + Testosterone
Number analyzed (Participants) | 11 | 7
picogram/milliliter | 13.35 (13.99) | 94.52 (200.92)

30. Secondary Outcome: Concentration of Cytokine Interleukin 10 (IL-10) in Blood as Measured by Immunoassay at 7 Weeks.
Description: as for outcome 29
Time Frame: 7 weeks
Population: Blood was collected for this outcome from only 18 subjects.
Measure: Mean (Standard Deviation); unit: picogram/milliliter
Arm/Group | Arm I: Standard of Care Therapy + Placebo Testosterone | Arm II: Standard of Care Therapy + Testosterone
Number analyzed (Participants) | 11 | 7
picogram/milliliter | 12.84 (13.25) | 82.46 (184.34)

31. Secondary Outcome: Concentration of Cytokine Interleukin 12 (IL-12) in Blood as Measured by Immunoassay at Baseline.
Description: Concentration of cytokine Interleukin 12 (IL-12) in blood as measured using Millipore Multiplex Human Cytokine Panel assay.
Time Frame: Baseline
Population: Blood was collected for this outcome from only 18 subjects.
Measure: Mean (Standard Deviation); unit: picogram/milliliter
Arm/Group | Arm I: Standard of Care Therapy + Placebo Testosterone | Arm II: Standard of Care Therapy + Testosterone
Number analyzed (Participants) | 11 | 7
picogram/milliliter | 3.94 (2.62) | 44.04 (91.34)

32. Secondary Outcome: Concentration of Cytokine Interleukin 12 (IL-12) in Blood as Measured by Immunoassay at 7 Weeks.
Description: as for outcome 31
Time Frame: 7 weeks
Population: Blood was collected for this outcome from only 18 subjects.
Measure: Mean (Standard Deviation); unit: picogram/milliliter
Arm/Group | Arm I: Standard of Care Therapy + Placebo Testosterone | Arm II: Standard of Care Therapy + Testosterone
Number analyzed (Participants) | 11 | 7
picogram/milliliter | 4.36 (2.40) | 28.36 (54.52)

33. Secondary Outcome: Concentration of Cytokine Interleukin 13 (IL-13) in Blood as Measured by Immunoassay at Baseline.
Description: Concentration of cytokine Interleukin 13 (IL-13) in blood as measured using Millipore Multiplex Human Cytokine Panel assay.
Time Frame: Baseline
Population: Blood was collected for this outcome from only 18 subjects.
Measure: Mean (Standard Deviation); unit: picogram/milliliter
Arm/Group | Arm I: Standard of Care Therapy + Placebo Testosterone | Arm II: Standard of Care Therapy + Testosterone
Number analyzed (Participants) | 11 | 7
picogram/milliliter | 2.50 (1.77) | 20.50 (39.60)

34. Secondary Outcome: Concentration of Cytokine Interleukin 13 (IL-13) in Blood as Measured by Immunoassay at 7 Weeks.
Description: as for outcome 33
Time Frame: 7 weeks
Population: Blood was collected for this outcome from only 18 subjects.
Measure: Mean (Standard Deviation); unit: picogram/milliliter
Arm/Group | Arm I: Standard of Care Therapy + Placebo Testosterone | Arm II: Standard of Care Therapy + Testosterone
Number analyzed (Participants) | 11 | 7
picogram/milliliter | 3.82 (3.42) | 17.95 (35.29)

35. Secondary Outcome: Concentration of Cytokine Tumor Necrosis Factor Alpha (TNFa) in Blood as Measured by Immunoassay at Baseline.
Description: Concentration of cytokine tumor necrosis factor alpha (TNFa) in blood as measured using Millipore Multiplex Human Cytokine Panel assay.
Time Frame: baseline
Population: Blood was collected for this outcome from only 18 subjects.
Measure: Mean (Standard Deviation); unit: picogram/milliliter
Arm/Group | Arm I: Standard of Care Therapy + Placebo Testosterone | Arm II: Standard of Care Therapy + Testosterone
Number analyzed (Participants) | 11 | 7
picogram/milliliter | 11.87 (3.02) | 13.88 (6.40)

36. Secondary Outcome: Concentration of Cytokine Tumor Necrosis Factor Alpha (TNFa) in Blood as Measured by Immunoassay at 7 Weeks.
Description: as for outcome 35
Time Frame: 7 weeks
Population: Blood was collected for this outcome from only 18 subjects.
Measure: Mean (Standard Deviation); unit: picogram/milliliter
Arm/Group | Arm I: Standard of Care Therapy + Placebo Testosterone | Arm II: Standard of Care Therapy + Testosterone
Number analyzed (Participants) | 11 | 7
picogram/milliliter | 33.52 (71.72) | 12.22 (6.02)

37. Secondary Outcome: Fat Mass as Measured by Dual Energy XRay Absorptiometry (DEXA) at Baseline
Description: Total Fat Mass as measured by dual energy xray absorptiometry at the baseline study visit
Time Frame: baseline
Population: 24 subjects were able to complete this outcome measure at the baseline study visit.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Arm I: Standard of Care Therapy + Placebo Testosterone | Arm II: Standard of Care Therapy + Testosterone
Number analyzed (Participants) | 12 | 12
grams | 20513.50 (13044.73) | 18227.33 (10470.48)

38. Secondary Outcome: Fat Mass as Measured by Dual Energy XRay Absorptiometry (DEXA) at 7 Weeks
Description: Total fat mass as measured by Dual Energy XRay Absorptiometry (DEXA) at the 7 week study visit.
Time Frame: 7 weeks
Population: 24 subjects began the study, 2 were dis-enrolled, 22 subjects finished the study. All 22 subjects completed this outcome measure at 7 weeks.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Arm I: Standard of Care Therapy + Placebo Testosterone | Arm II: Standard of Care Therapy + Testosterone
Number analyzed (Participants) | 12 | 10
grams | 17616.58 (12513.32) | 16776.60 (10989.56)

39. Secondary Outcome: Quality of Life Measurement as Measured by Medical Outcome Study - Short Form 36 at Baseline
Description: The Medical Outcome Study - Short Form 36 (MOS-SF-36) is a questionnaire developed by RAND Health to measure patient self-reported quality of life. Data presented is a subset of the questionnaire, Scale of General Health. The range for the subset presented (General Health) is 0 - 100, with 100 being better perceived health and 0 being worst perceived health. The national average of the MOS-36 General Health Subscale is reported as 56.99.
Time Frame: baseline
Population: 20 subjects completed this questionnaire at this time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I: Standard of Care Therapy + Placebo Testosterone | Arm II: Standard of Care Therapy + Testosterone
Number analyzed (Participants) | 11 | 9
units on a scale | 47.73 (27.87) | 52.22 (23.60)

40. Secondary Outcome: Quality of Life Measurement as Measured by Medical Outcome Study - Short Form 36 at 7 Weeks
Description: as for outcome 39
Time Frame: 7 weeks
Population: 21 subjects completed this questionnaire at this time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Arm I: Standard of Care Therapy + Placebo Testosterone | Arm II: Standard of Care Therapy + Testosterone
Number analyzed (Participants) | 11 | 10
Units on a scale | 52.73 (22.73) | 46.50 (14.54)

41. Secondary Outcome: Personal Perception of Fatigue as Measured by Multidimensional Fatigue Symptom Inventory - Short Form at Baseline
Description: Multidimensional Fatigue Symptom Inventory Short Form (MFSI-SF) from the Moffitt Cancer Center, University of South Florida The MFSI-SF is a 30 question assessment designed to assess the principal manifestations of fatigue.
  There 5 subscales used to calculate a total score. The subscales are: General Fatigue, Physical Fatigue, Emotional Fatigue, Mental Fatigue, and Vigor (an estimate of the patient's energy level). The total score is calculated with the equation: (general + physical + emotional + mental) - vigor = total score.
  The range of the total score is -24 to 96, with the higher the number meaning more fatigue.
Time Frame: Baseline
Population: 21 subjects completed this questionnaire at this time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Arm I: Standard of Care Therapy + Placebo Testosterone | Arm II: Standard of Care Therapy + Testosterone
Number analyzed (Participants) | 11 | 10
Units on a scale | 12.73 (25.48) | 21.40 (21.27)

42. Secondary Outcome: Personal Perceptual Fatigue Measured by Multidimensional Fatigue Symptom Inventory at 7 Weeks
Description: as for outcome 41
Time Frame: 7 weeks
Population: 20 subjects completed this questionnaire at this time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Arm I: Standard of Care Therapy + Placebo Testosterone | Arm II: Standard of Care Therapy + Testosterone
Number analyzed (Participants) | 11 | 9
Units on a scale | 18.73 (24.18) | 26.11 (19.73)

43. Secondary Outcome: Mood Measured by Profile of Mood States at Baseline
Description: Profile of Mood States (POMS) is a questionnaire by MultiHealth Systems, that measures mood. In this 65 item questionnaire, subjects are asked to rate their feelings toward a statement from 0-4, with 0 being "not at all' and 4 being "extremely". There are 6 subscales which include, tension-anxiety, depression, anger-hostility, vigor, fatigue, and confusion. To calculate the total mood disturbance, which is what is reported here, the subscales tension-anxiety, depression, anger-hostility, fatigue and confusion are summed and vigor is subtracted. The scale range for total mood disturbance is 200 (worst) to -32 (best).
Time Frame: baseline
Population: 22 subjects completed this questionnaire at this time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I: Standard of Care Therapy + Placebo Testosterone | Arm II: Standard of Care Therapy + Testosterone
Number analyzed (Participants) | 11 | 11
units on a scale | 30.73 (50.67) | 32.55 (23.74)

44. Secondary Outcome: Mood as Measured by Profile of Mood States at 7 Weeks
Description: as for outcome 43
Time Frame: 7 weeks
Population: 20 subjects completed this questionnaire at this time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Arm I: Standard of Care Therapy + Placebo Testosterone | Arm II: Standard of Care Therapy + Testosterone
Number analyzed (Participants) | 11 | 9
Units on a scale | 28.82 (44.18) | 35.78 (36.81)

45. Secondary Outcome: Quality of Life as Measured by Functional Assessment of Cancer Therapy - General Questionnaire at Baseline
Description: Functional Assessment of Cancer Therapy - General (FACT-G) is a patient-reported questionnaire of quality of life. The 27 item questionnaire is separated into 4 subscales, physical well-being, social/family well-being, emotional well-being, functional well-being. These subscales are summed to calculate total score. The range for FACT-G is 0 (worst quality of life) to 108 (best quality of life).
Time Frame: Baseline
Population: 19 subjects completed this questionnaire at this time point.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Arm I: Standard of Care Therapy + Placebo Testosterone | Arm II: Standard of Care Therapy + Testosterone
Number analyzed (Participants) | 9 | 10
scores on a scale | 18.83 (3.50) | 30.48 (31.63)

46. Secondary Outcome: Quality of Life as Measured by Functional Assessment of Cancer Therapy - General Questionnaire at 7 Weeks
Description: as for outcome 45
Time Frame: 7 weeks
Population: 20 subjects completed this questionnaire at this time point.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Arm I: Standard of Care Therapy + Placebo Testosterone | Arm II: Standard of Care Therapy + Testosterone
Number analyzed (Participants) | 9 | 10
scores on a scale | 20.11 (4.04) | 24.97 (20.18)

47. Secondary Outcome: 1-year Survival
Description: Number of participants who survived one year post study.
Time Frame: 1 year post study
Population: 12 subjects started each group. 2 subjects withdrew after baseline from the testosterone group.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I: Standard of Care Therapy + Placebo Testosterone | Arm II: Standard of Care Therapy + Testosterone
Number analyzed (Participants) | 12 | 10
Participants | 7 | 6

ADVERSE EVENTS:
Time Frame: 7 weeks
Arm/Group | Arm I: Standard of Care Therapy + Placebo Testosterone | Arm II: Standard of Care Therapy + Testosterone
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 6/12 | 6/12
Other Adverse Events (participants affected / at risk) | 6/12 | 3/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I: Standard of Care Therapy + Placebo Testosterone (N=12) | Arm II: Standard of Care Therapy + Testosterone (N=12)
Anemia Requiring Tranfusion (Blood and lymphatic system disorders) | 5 (9) | 3 (6)
Duodenal Ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) — Duodenal Ulcer that caused anemia and required a blood tranfusion
Cerebrovascular Accident (Vascular disorders) | 1 (1) | 0 (0)
Anaphylactic shock (General disorders) | 1 (1) | 0 (0) — Anaphylactic shock to chemotherapy agen
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Sycope (General disorders) | 0 (0) | 1 (1) — Syncope resulting in a fall with broken arm
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I: Standard of Care Therapy + Placebo Testosterone (N=12) | Arm II: Standard of Care Therapy + Testosterone (N=12)
Dysphagia (General disorders) | 1 (1) | 0 (0)
Fever (Infections and infestations) | 2 (2) | 0 (0) — Fever requiring anitbiotics
Neutropenic Fever (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 4 (5) | 2 (2)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Altered Mental State (Psychiatric disorders) | 1 (1) | 0 (0)
Hyponatremia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Vesicovaginal Fistula (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Metastatic Bowel Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No